CLINICAL TRIAL: NCT01821989
Title: Oral Lactoferrin Supplementation for Prevention of Sepsis in Preterm Neonate.
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mooselmokadem (Other)
Responsible Party: Principal Investigator, Mostafa El-Mokadem, neonatologist, Mooselmokadem
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: moos80
Record Dates: First submitted 2013-03-27; First posted 2013-04-01 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Neonatal Sepsis
MeSH Terms: conditions — Neonatal Sepsis | interventions — Lactoferrin

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor

ARMS (3):
- Low Dose (Active Comparator): Lactoferrin,dose of 100 mg/day.
  Interventions: Dietary Supplement: Lactoferrin
- High Dose (Experimental): Lactoferrin, dose of 150 mg/kg/ twice daily.
  Interventions: Dietary Supplement: Lactoferrin
- Control (Placebo Comparator): Receive placebo in form of distilled water.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactoferrin — dose of 100 mg/day
  Arms: Low Dose
Dietary Supplement: Lactoferrin — dose of 150 mg/kg/ twice daily
  Arms: High Dose
Dietary Supplement: Placebo — in form of distilled water
  Arms: Control

SUMMARY:
Hypothesis:

Orally ingested lactoferrin has effects on promotion of growth and differentiation of the immature gut; also it has immunomodulatory properties, so it will prevent serious infections in preterm infants.

The aim of the study is to:

* Evaluate the effectiveness of oral lactoferrin in prevention of neonatal sepsis.
* Compare two dose regiment of lactoferrin supplementation.
* Study effect of lactoferrin supplementation on serum iron stores.

It is a prospective, randomized, double blind, placebo-controlled study, it will include 180 preterm neonates admitted to the Neonatal Intensive Care Units of of Ain Shams University Hospitals and Manshiet El Bakry Hospital.

•Group A: Who will receive oral lactoferrin supplementation in a dose of 100 mg/day.

•Group B: Who will receive oral lactoferrin supplementation in a dose of 150 mg/kg/ twice daily.

•Group C (Controls): Who match the subjected neonates, will receive placebo in form of distilled water.

ELIGIBILITY:
Inclusion Criteria:

1. Neonates with a birth weight between 500g and 2500g.
2. Neonates with a ≤ 36 weeks of gestation counting from the first day of the Last Menstrual Period.
3. Preterm neonates born in, or referred to the Neonatal Intensive Care Units of one of the participating hospitals in the first 48 hours of life.

Exclusion Criteria:

1. Neonates with underlying gastrointestinal problems that prevent oral intake.
2. Neonates with predisposing conditions that profoundly affect growth and development (chromosomal abnormalities, structural brain anomalies, severe congenital abnormalities).
3. Neonates with a family background of cow milk allergy.
4. Neonates who will not have the chance to complete the study time (who will be referred to another hospitals).
5. Neonates whose parents decline to participate.
6. Neonates with early onset sepsis.

Max Age: 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2013-06; Primary Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Blood culture | 2 years

SECONDARY OUTCOMES:
Complete blood count with differential leucocytic count. | 2 years

OTHER OUTCOMES:
C reactive protein quantitative assay | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Abassia, Egypt